CLINICAL TRIAL: NCT06332677
Title: Targeting the Epigenetic Regulators Suv420h1/2 in Hepatocytes to Treat Nonalcoholic Fatty Liver Disease
Brief Title: Target of Suv420h1/2 in Hepatocytes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Valenti:, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TERS
Record Dates: First submitted 2024-03-08; First posted 2024-03-27 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: NAFLD
Keywords: epigenetic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: study the cellular and molecular mechanisms of correlation between the SUV420H1/H2 methyltransferase and the progression of liver damage in mice (San Raffaele Institute) and to confirm these findings in human samples and in vitro 3D liver models.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the main genes and expression by comparing the transcriptomic lipidomic profile (Experimental): To identify the main genes and pathways differentially expressed and the main factors associ- ated with SUV420H1/H2 expression by comparing the transcriptomic and lipidomic profile of indi- viduals with low hepatic SUV420H1/H2 mRNA expression levels (lowest expression quartile) to that from individuals with high expression levels (top quartile).
  In order to evaluate the role of SUV420H1/H2 in the regulation of gene expression in NAFLD pa- tients, we will exploit already available transcriptomic and lipidomic data by analyzing the gene ex- pression databases deriving from ongoing studies conducted at the Fondazione and by the PI of the Catanzaro collaborating centre. Data have been generated from liver and visceral adipose biopsy of obese individuals at high risk of developing NASH (SERENA Study at Fondazione, and MAFALDA Study, coordinated by prof Stefano Romeo, PI of the Università Magna Graecia Catanzaro).
  Interventions: Diagnostic Test: the main genes and expression by comparing the transcriptomic lipidomic profile

INTERVENTIONS:
Diagnostic Test: the main genes and expression by comparing the transcriptomic lipidomic profile — To identify the main genes and pathways differentially expressed and the main factors associ- ated in order to evaluate the role of SUV420H1/H2

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is globally the leading cause of liver disease and frequently progresses to cirrhosis and liver cancer. The identification of effective drugs is the main unmet clinical need. Changes in liver histones methylation accompanies the development and progression of NAFLD. Our preliminary data demonstrate that inactivation of the methyltransferases SUV420H1/2 in hepatocytes protects mice against NAFLD. In this project we propose to examine the relevance of these findings by evaluating the impact of genetic deletion of hepatic SUV420H1/2 in mice fed a steatogenic diet. To further evaluate the potential for clinical translation of these results, we will next 1) evaluate the expression of SUV420H1/2 in human liver transcriptomic data and 2) analyze the impact of genetic variations on disease outcomes in population-based cohorts; 3) test an innovative therapeutic approach based on hepatocyte-targeted antisense oligonucleotides downregulating SUV420H1/2 in human liver organoids/assembloids.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD), the leading cause of liver damage worldwide, is characterized by liver fat accumulation and association with insulin resistance, and frequently progresses to steatohepatitis (NASH), ultimately leading to cirrhosis and liver cancer.

NAFLD/NASH is becoming globally a leading cause of liver-related morbidity and mortality and by altering liver function contributes more widely to the burden of cardiometabolic, renal and neoplastic diseases. In the presence of concomitant hepatotoxic factors such as in particular atrisk alcohol intake and some medications (defined in this case as metabolic dysfunction associated fatty liver disease or MAFLD) synergizes with them representing a major driver of liver disease progression. However, for those with advanced disease or who cannot successfully change their diet and lifestyle, no effective treatment is yet available to prevent or treat this condition, which is therefore projected to become a major public health threat in the next decade. Although understanding the mechanisms of NAFLD development and progression is essential for its prevention/treatment, molecular players involved in its progression are poorly defined. Recently, an epigenetic component is recognized in this disorder and the histone methyltransferases SUV420H1/2 are promising candidates for this function. Multiple evidences connect lipid and iron metabolism in the hepatocyte: 1) Genome Wide Association Studies (GWAS) in human populations showed an overlap of loci affecting iron and lipid metabolism, and excess iron in hepatocytes favors dyslipidemia and NAFLD; 2) upregulation of the liver hormone hepcidin, under the control by the BMP-SMAD pathway, is protective against NAFLD-NASH. Interestingly, a GWAS performed in mouse strains kept on high-iron diet identified a shared association between liver iron and triglyceride levels at a region of chromosome 7 encompassing the histone methyltransferase Suv420h2. Our preliminary data show that mice with Suv420h inactivation in adipose tissue are resistant to diet-induced liver steatosis due to increased PPAR signaling. Since mice with liver BMP-SMAD pathway upregulation showed Suv420h downregulation, we hypothesize that the protective effect of increased hepatocyte BMP-SMAD signaling on NAFLD development is due to Suv420h. In agreement, Suv420h inactivation in hepatocytes counteracts diet-induced NAFLD, as highlighted by our preliminary results.

The present study is part of the RF project (Ricerca Finalizzata) - Project code: RF-2021-12373889 funded by the grant call of the Ministery of Health (2020-2021). In the attached project we proposed 3 different aims:

* To characterize the disease progression in Suv420h1/2-liver conditional KO mice and to identify
* To examine the impact of SUV420H1/2 genetic, epigenetic and transcriptional variability on clinical outcomes for the identification of novel biomarkers of NAFLD-NASH.
* To propose and test an innovative therapeutic approach based on hepatocyte-targeted antisense oligonucleotides (ASOs) against Suv420h1/2 in preclinical models in mice and in human liver organoids and assembloids. The present clinical study protocol will focus on the clinical aspects and procedures that will regard an intervention on data and sample of clinical cohorts. Further details about the analyses conducted in animal models, for which a specific Authorization has been requested, can be found in the attached project.

ELIGIBILITY:
Inclusion Criteria:

We will analyse data and samples from subjects with the following criteria:

* Subjects aged>18;
* Subjects who have already given their consent to genetic analysis and whose samples and data have already been collected as part of the SERENA, REASON and MAFALDA studies;
* Subjects who have given their consent to participate in this study.

In particular, subjects with the following characteristics were included respectively:

* in the SERENA study:

  1. Diagnosis of NAFLD
  2. Age between 45 and 75 years old
  3. Any of the following criteria:

     1. F3-F4 fibrosis, determined histologically, or by non-invasive techniques, or evidence of cirrhosis deriving from biochemical tests or imaging methods;
     2. Family history of related first-degree primary liver cancer, or carrier status of rare mutations associated with the development of HCC (such as mutations in APOB and TERT)
     3. Male patient with type 2 diabetes or obesity carrying at least three genetic variants in PNPLA3, TM6SF2, MBOAT7.
* in the REASON study:

Patients aged>18, who have given their consent to participate in the study, who underwent the fol- lowing procedures:

* liver biopsy for suspected non-alcoholic steatohepatitis (NASH) at the time of diagnosis;
* liver resection for hepatocarcinoma, other liver lesions (including secondaries from other neo- plasms and benign focal lesions, which will allow obtaining healthy starting liver tissue), biopsies of whole liver explants obtained at the time of liver transplantation AND cholecystectomies.
* In the MAFALDA study:

Patients undergoing bariatric surgery for grade 3 obesity (BMI ≥40 Kg/m2) or grade 2 obesity plus:

* metabolic comorbidities (uncontrolled hypertension, diabetes, dyslipidemia);
* lack of contraindication to surgery (e.g. advanced liver disease with portal hypertension);
* willingness to sign an informed consent.

Exclusion Criteria:

* Individuals not reporting one of the inclusion criteria listed above or reporting at-risk alcohol intake (>30/20 g/day in M/F), viral and autoimmune hepatitis or other causes of liver disease will be ex- cluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
the main genes and expression by comparing the transcriptomic lipidomic profile | up to 30 mounths
  The primary aim is the identification of biological pathways differentially ex- pressed in NAFLD individuals.
  Considering the large number of individuals with severe liver disease in the NAFLD PERSPECTIVE and MAFALDA cohorts (n= 500) and the large size of UKBB population-based cohort (n=350,000 for common variants and n=200,000 for rare variants), for variants with a minor allele frequency (MAF) >0.01, we estimated that the study has a power >80% to detect six-fold difference in the risk of severe NAFLD in the PERSPECTIVE/MAFALDA, a 1.8% difference in the NAFLD prevalence (UK Biobank), and 4.4% difference in the liver fat content as measured by PDFF (UK Biobank) between carriers and non-carriers (Aim A and B).
the main genes and expression by comparing the transcriptomic lipidomic profile | up to 30 mounths
  The identification of a correlation between genotype influencing the SUV420H1/2 pathway and NAFLD phenotype.
  Reduction of intracellular fat accumulation, collagen accumulation and inflammation in terms of TNFalpha mRNA expression levels.
  In case of positive results from SUV420H1/H2 downregulation by antisense technology, both in mouse models than in human liver organoids and assembloids, we will submit a patent request for the human anti-SUV420H1-H2 ASO for the treatment of steatohepatitis (Fondazione IRCCS Ca' Granda and San Raffaele Institute).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT06332677/Prot_SAP_000.pdf